CLINICAL TRIAL: NCT04065412
Title: Modified Laryngeal Handshake Technique for Locating the Cricothyroid Membrane
Brief Title: Modified Laryngeal Handshake Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2019208
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Airway Complication of Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional laryngeal handshake technique (Active Comparator): The conventional laryngeal handshake technique is performed to localize the cricothyroid membrane
  Interventions: Procedure: Conventional laryngeal handshake technique
- Modified laryngeal handshake technique (Experimental): The modified laryngeal handshake is performed to localize the cricothyroid membrane
  Interventions: Procedure: Modified laryngeal handshake technique

INTERVENTIONS:
Procedure: Conventional laryngeal handshake technique — The conventional laryngeal handshake technique is performed with the non-dominant hand, identifying the hyoid bone and thyroid laminae, stabilizing the larynx between thumb and middle finger, and moving down the neck to palpate the cricothyroid membrane with the index finger.
  Arms: Conventional laryngeal handshake technique
Procedure: Modified laryngeal handshake technique — The modified laryngeal handshake is performed with the non-dominant hand, stabilizing the trachea between thumb and middle finger from the suprasternal notch and moving up the neck to palate the cricoid cartilage and cricothyroid membrane with the index finger.
  Arms: Modified laryngeal handshake technique

SUMMARY:
In this study, we compare the conventional laryngeal handshake technique and modified laryngeal handshake technique for locating the cricothyroid membrane in terms of accuracy and speed. The conventional laryngeal handshake technique is performed with the non-dominant hand, identifying the hyoid bone and thyroid laminae, stabilizing the larynx between thumb and middle finger, and moving down the neck to palpate the cricothyroid membrane with the index finger.

The modified laryngeal handshake is performed with the non-dominant hand, stabilizing the trachea between thumb and middle finger from the suprasternal notch and moving up the neck to palate the cricoid cartilage and cricothyroid membrane with the index finger.

ELIGIBILITY:
Inclusion Criteria:

* Patients who would be scheduled elective surgery under general anesthesia

Exclusion Criteria:

* Diseases or anatomical abnormalities in the neck or larynx
* History of neck surgery

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
The accuracy to localize the cricothyoid membrane | 1 minute after identifying the cricothyroid membrane using the conventional or modified laryngeal handshake technique
  The accuracy of the cricothyroid membrane identified by the conventional and modified handshake techniques are evaluated.

SECONDARY OUTCOMES:
The accuracy to localize the midline of the neck | through the identification of cricothyroid membrane, an average of 5 minutes
  The accuracy of the midline of the neck identified by the conventional and modified handshake techniques are evaluated.
The vertical and horizontal distances between the actual and perceived cricothyroid membrane | through the identification of cricothyroid membrane, an average of 5 minutes
  The vertical and horizontal distances between the actual and perceived cricothyroid membrane using the conventional and modified handshake techniques are evaluated.
Time to localize the cricothyroid membrane | through the identification of cricothyroid membrane, an average of 5 minutes
  The time taken to identify the cricothyroid membrane is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Chang JE, Kim H, Won D, Lee JM, Kim TK, Min SW, Hwang JY. Comparison of the Conventional Downward and Modified Upward Laryngeal Handshake Techniques to Identify the Cricothyroid Membrane: A Randomized, Comparative Study. Anesth Analg. 2021 Nov 1;133(5):1288-1295. doi: 10.1213/ANE.0000000000005744. PMID 34517392